CLINICAL TRIAL: NCT06100991
Title: CorEvitas Generalized Pustular Psoriasis (GPP) Drug Safety and Effectiveness Registry
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: GPP-510
Record Dates: First submitted 2023-10-03; First posted 2023-10-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Generalized Pustular Psoriasis (GPP): Pts presenting to enrolling sites across the North America are invited to enroll if eligible

SUMMARY:
Prospective, observational registry for subjects with GPP under the care of a dermatology investigator.Approximately 200 subjects and 75 clinical sites in North America will be recruited to participate with no defined upper limit for either target

DETAILED DESCRIPTION:
The objective of the registry is to obtain information on the treatment patterns, disease activity progression, and the development of comorbidities and adverse events in a cohort of patients with GPP. Data collected will be used to better characterize the natural history and longitudinal trajectory of the disease. This will be done through the standardized data collection including validated patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization patterns. Personal information is also collected from each consenting registry subject allowing for linkages to other public or private clinical and administrative databases, as well as to databases maintained by organizations focused on the care and treatment of GPP for the purposes of clinical, market, or outcomes research.

This provides an opportunity to evaluate other aspects of the disease and its treatment, including but not limited to clinical and drug cost-effectiveness, health care resource utilization, and subject adherence.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet all the following criteria to participate in the registry:

  1. Has been diagnosed with GPP by a dermatologist or a qualified dermatology practitioner.
  2. Is at least 18 years of age and has attained the legal age for consent to procedures involved in the research, under the applicable law of the jurisdiction in which the research is being conducted.
  3. Is willing to provide consent for participation in the registry.
  4. Is willing to provide Personal Information

Exclusion Criteria:

* Any of the following would exclude the subject from participating in the registry:

  1. Is participating or planning to participate in a blinded clinical trial evaluating a systemic agent for the treatment or prevention of flares related to GPP.
  2. Is enrolled in another CorEvitas registry for a dermatological condition. Subjects enrolled in another CorEvitas registry must be exited to be eligible for enrollment into the GPP Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are enrolled in the GPP Registry during regularly scheduled office visits. Selected dermatologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure:GPP epidemiology and Presentation | Through study completion, an average of 10 years
  The major clinical outcomes include an assessment of the epidemiology of GPP; to better understand the presentation and natural history.
GPP management, and outcomes | Through study completion, an average of 10 years
  The major clinical outcome include an assessment of the epidemiology of GPP; to better understand the management and outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://corevitas.com/